CLINICAL TRIAL: NCT03800810
Title: Potency of Allogenic Umbilical Cord Mesenchymal Stem Cells for Osteoarthritis Management
Brief Title: Implantation of Allogenic Mesenchymal Stem Cell From Umbilical Cord Blood for Osteoarthritis Management
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Ismail Hadisoebroto Dilogo, Consultant, Department of Orthopaedics and Traumatology, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ISMMSCOA
Record Dates: First submitted 2018-07-02; First posted 2019-01-11 (Actual); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Osteoarthritis, Knee
Keywords: Osteoarthritis; Mesenchymal Stem Cells; Umbilical Cord
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — Hyaluronic Acid; Human Growth Hormone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Control (Experimental): Week 1: Intraarticular injection of 2 ml hyaluronic acid (Synvisc-One® Hylan G-F 20, Sanofi-Aventis) Week 2: Intraarticular injection of 2 ml hyaluronic acid (Synvisc-One® Hylan G-F 20, Sanofi-Aventis) Week 3: Intraarticular injection of 2 ml hyaluronic acid (Synvisc-One® Hylan G-F 20, Sanofi-Aventis)
  Interventions: Drug: Hyaluronic Acid
- Intervention 1 (Experimental): Week 1: Intraarticular injection of 10x10^6 unit of umbilical cord mesenchymal stem cells in 2 ml conditioned medium, 2 ml hyaluronic acid (Synvisc-One® Hylan G-F 20, Sanofi-Aventis) Week 2: Intraarticular injection of 2 ml hyaluronic acid (Synvisc-One® Hylan G-F 20, Sanofi-Aventis), 8 IU recombinant human somatropin (Novell-Eutropin®, Novell Pharmaceutical Laboratories) Week 3: Intraarticular injection of 2 ml hyaluronic acid (Synvisc-One® Hylan G-F 20, Sanofi-Aventis), 8 IU recombinant human somatropin (Novell-Eutropin®, Novell Pharmaceutical Laboratories)
  Interventions: Drug: Hyaluronic Acid; Biological: Umbilical Cord Mesenchymal Stem Cell; Biological: Recombinant Human Somatropin
- Intervention 2 (Experimental): Week 1: Intraarticular injection of 10x10^6 unit of umbilical cord mesenchymal stem cells in 2 ml conditioned medium, 2 ml hyaluronic acid (Synvisc-One® Hylan G-F 20, Sanofi-Aventis) Week 2: Intraarticular injection of 2 ml hyaluronic acid (Synvisc-One® Hylan G-F 20, Sanofi-Aventis) Week 3: Intraarticular injection of 2 ml hyaluronic acid (Synvisc-One® Hylan G-F 20, Sanofi-Aventis)
  Interventions: Drug: Hyaluronic Acid; Biological: Umbilical Cord Mesenchymal Stem Cell
- Intervention 3 (Experimental): Week 1: Intraarticular injection of 10x10^6 unit of umbilical cord mesenchymal stem cells in 2 ml conditioned medium, 2 ml hyaluronic acid (Synvisc-One® Hylan G-F 20, Sanofi-Aventis) Week 2: Intraarticular injection of 2 ml hyaluronic acid (Synvisc-One® Hylan G-F 20, Sanofi-Aventis), 8 IU recombinant human somatropin (Novell-Eutropin®, Novell Pharmaceutical Laboratories) Week 3: Intraarticular injection of 2 ml hyaluronic acid (Synvisc-One® Hylan G-F 20, Sanofi-Aventis), 8 IU recombinant human somatropin (Novell-Eutropin®, Novell Pharmaceutical Laboratories)
  Interventions: Drug: Hyaluronic Acid; Biological: Recombinant Human Somatropin

INTERVENTIONS:
Drug: Hyaluronic Acid
  Other Names: Hyaluronan
Biological: Umbilical Cord Mesenchymal Stem Cell
  Arms: Intervention 1; Intervention 2
Biological: Recombinant Human Somatropin
  Arms: Intervention 1; Intervention 3

SUMMARY:
Prevalence of osteoarthritis increases every year, as a chronic and progressive disease. Osteoarthritis also gives many negative impacts in socio-economic life. Current management of osteoarthritis only aimed to relieve pain but not to resolve the degeneration of cartilage. Mesenchymal stem cell is one kind of adult stem cell that has potency in tissue engineering. Sources of mesenchymal stem cell are bone marrow, adipose tissue and umbilical cord. Researchers want to explore the potential of umbilical cord as the source of allogeneic MSC, because the gaining process of MSC is not invasive. Some countries have started some In vitro studies, Animal studies, and human research, but in Indonesia the study of mesenchymal stem cell implantation from umbilical cord in genu osteoarthritis management has not been reported. This study will be held into two years in Cipto Mangunkusumo Hospital and include 9 participants minimally. The researcher also compares the efficacy and safety of MSC implantation from umbilical cord applied to genu osteoarthritis with synovial artificial and recombinant human growth hormone therapy.

DETAILED DESCRIPTION:
This study is experimental clinical, randomized control trial. This study estimated time would be 24 months, from May 2016 until May 2018. Samples are obtained consecutively from all source population that meet criteria. This study divide the samples into three groups, synovial artificial group, MSC and synovial artificial combination group; MSC, Synovial, and recombinant human growth hormone group. The number of samples in each group is three.

Subject Criteria Inclusion Criteria for MSC Donor from Umbilical Cord:

Umbilical cord are collected from elective caesarean section from a fullterm pregnancies without any complication and free from HIV, Hepatitis B, C, D virus, Cytomegalovirus, Rubella Virus, and free from fungal and bacterial contamination.

Recipient inclusion criteria of osteoarthritis samples are patients aged 30-80 years old, based on genu X-ray examination and Kellgren-Lawrence grading is I, II, and III, or KL grade III with corrective osteotomy, minimal Visual Analog Scale = 2 (0-10), unresponsive with pharmacological therapy, and also sign up the informed consent.

Recipient exclusion criteria are Osteoarthritis KL grade IV, and secondary osteoarthritis due to trauma, infection, rheumatoid arthritis, congenital diseases, and autoimmune diseases, hypersensitivity of hyaluronan product, cancer, pregnant women.

Drop Out Criteria patients are ruled out from this study while the research are held or they undergo another treatment that are not related to this study. All drop out subjects could get another treatment.

Informed consent all of subjects must be filled and signed up before ruled in this study.

As soon as after delivery, umbilical cord is collected and processed in sterile specimen 0,9% NaCl at 4oC during 8 hours. The umbilical cord transported to the laboratory and cultured in GMP lab, at UPTTK Sel Punca Cipto Mangunkusumo Hospital. Cellular viability and proliferation are evaluated after cell characterization test by flowcytometer.

Sterility test are done three times to ensure cellular sterility. Subjects are positioned in supine position, site of injection are determined by the operator. Injection from superolateral or superomedial in extension knee position, injection from anterolateral or anteromedial in flexion knee position. Aseptic and antiseptic in site of injection use povidone iodine 3 times, then swab by alcohol. Local anesthetic by lidocaine 1% is injected subcutaneously.

Monitoring at the site of injection encompass allergic reaction, pain, and swelling. Patients are approached to be followed up every three months, in 1st ,3rd ,6th ,12th month, for clinical examination, VAS, IKDC and WOMAC Score. Cartigram MRI are evaluated every six month, in 6th and 12th month.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 30-80 years old
* Kellgren-Lawrence grade I, II, and III, or KL grade III with corrective osteotomy according to knee x-ray examination
* Minimal VAS: 2
* Unresponsive with pharmacological therapy
* Signed the informed consent

Exclusion Criteria:

* Osteoarthritis KL grade IV
* Secondary osteoarthritis due to trauma, infection, rheumatoid arthritis, congenital diseases, autoimmune diseases
* Hypersensitivity to hyaluronic acid
* Malignancies (Previously or currently diagnosed)
* Pregnancy

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2015-05; Primary Completion 2019-05 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
Cartilage T2 map score | 6 months
  MRI examination of the knee with additional T2 mapping software CartiGram (GE Healthcare, USA). T2 map sequence are obtained from the medial and lateral aspect of both femoral and tibial cartilage.
IKDC score | 3 months
  Subjective assessment of knee function using the International Knee Documentation Committee Subjective Knee Evaluation form.
  Scale ranges from 1 to 100, higher value indicates higher function.
WOMAC score | 3 months
  Subjective assessment of knee function using the the Western Ontario and McMaster Universities Osteoarthritis Index.
  Scale ranges from 100% to 1%, lower value indicates higher function.
VAS score | 3 months
  VAS score is used to assess knee pain experienced by subjects.

CONTACTS AND LOCATIONS:
Locations (1):
- Universitas Indonesia, Jakarta Pusat, Jakarta Special Capital Region, Indonesia

IPD SHARING:
Plan to Share IPD: Yes
Name Gender Contact Address Sign up

REFERENCES:
- [Background] Solomon L, Warwic DJ, Nagayam S. Osteoarthritis. In : Apple's System if Orthopaedics and Fractures 8th Edition.oxford University Press. New York : 2001. P 77-90
- [Background] Singh A, Goel SC, Gupta KK, Kumar M, Arun GR, Patil H, Kumaraswamy V, Jha S. The role of stem cells in osteoarthritis: An experimental study in rabbits. Bone Joint Res. 2014 Feb 13;3(2):32-7. doi: 10.1302/2046-3758.32.2000187. Print 2014. PMID 24526748
- [Background] Tsai SY, Huang YC, Chueh LL, Yeh LS, Lin CS. Intra-articular transplantation of porcine adipose-derived stem cells for the treatment of canine osteoarthritis: A pilot study. World J Transplant. 2014 Sep 24;4(3):196-205. doi: 10.5500/wjt.v4.i3.196. PMID 25346893
- [Background] Kim SB, Kwon DR, Kwak H, Shin YB, Han HJ, Lee JH, Choi SH. Additive effects of intra-articular injection of growth hormone and hyaluronic acid in rabbit model of collagenase-induced osteoarthritis. J Korean Med Sci. 2010 May;25(5):776-80. doi: 10.3346/jkms.2010.25.5.776. Epub 2010 Apr 16. PMID 20436717
- [Background] Vangsness CT Jr, Farr J 2nd, Boyd J, Dellaero DT, Mills CR, LeRoux-Williams M. Adult human mesenchymal stem cells delivered via intra-articular injection to the knee following partial medial meniscectomy: a randomized, double-blind, controlled study. J Bone Joint Surg Am. 2014 Jan 15;96(2):90-8. doi: 10.2106/JBJS.M.00058. PMID 24430407
- [Background] Dart AJ, Little CB, Hughes CE, Chu O, Dowling BA, Hodgson DR, Rose RJ, Johnson KA. Recombinant equine growth hormone administration: effects on synovial fluid biomarkers and cartilage metabolism in horses. Equine Vet J. 2003 May;35(3):302-7. doi: 10.2746/042516403776148165. PMID 12755435
- [Background] White DK, Keysor JJ, Lavalley MP, Lewis CE, Torner JC, Nevitt MC, Felson DT. Clinically important improvement in function is common in people with or at high risk of knee OA: the MOST study. J Rheumatol. 2010 Jun;37(6):1244-51. doi: 10.3899/jrheum.090989. Epub 2010 Apr 15. PMID 20395640
- [Background] Raynauld JP, Torrance GW, Band PA, Goldsmith CH, Tugwell P, Walker V, Schultz M, Bellamy N; Canadian Knee OA Study Group. A prospective, randomized, pragmatic, health outcomes trial evaluating the incorporation of hylan G-F 20 into the treatment paradigm for patients with knee osteoarthritis (Part 1 of 2): clinical results. Osteoarthritis Cartilage. 2002 Jul;10(7):506-17. doi: 10.1053/joca.2002.0798. PMID 12127830
- [Background] Higgins LD, Taylor MK, Park D, Ghodadra N, Marchant M, Pietrobon R, Cook C; International Knee Documentation Committee. Reliability and validity of the International Knee Documentation Committee (IKDC) Subjective Knee Form. Joint Bone Spine. 2007 Dec;74(6):594-9. doi: 10.1016/j.jbspin.2007.01.036. Epub 2007 Aug 6. PMID 17888709
- [Background] Sinusas K. Osteoarthritis: diagnosis and treatment. Am Fam Physician. 2012 Jan 1;85(1):49-56. PMID 22230308
- See also: Lozada, CJ. Et al. Osteoarthritis — http://emedicine.medscape.com/article/330487-overview
- See also: Hamami, MB. Growth Hormone — http://emedicine.medscape.com/article/2089136-overview
- See also: Anonimous. WOMAC index — https://www.rheumatology.org/Practice/Clinical/Clinicianresearchers/Outcomes_Instrumentation/Western_Ontario_and_McMaster_Universities_Osteoarthritis_Index_%28WOMAC%29/